CLINICAL TRIAL: NCT02426073
Title: Pilot Observational Study to Characterize Glucose Metabolism, Muscle Mass/Function and Inflammatory Profile in Elderly Individuals
Brief Title: Glucose Metabolism, Muscle Mass/Function and Inflammation in the Elderly
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: University of Rome Tor Vergata (Other); Fondazione Roma (Unknown)
Responsible Party: Principal Investigator, Giaccari Andrea, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5312/15
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Sarcopenia; Diabetes Mellitus
Keywords: Inflammaging
MeSH Terms: conditions — Sarcopenia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- HE: Healthy elderlies
- DM: Elderlies with type 2 diabetes
- SA: Elderlies with sarcopenia
- DS: Elderlies with both type 2 diabetes and sarcopenia

SUMMARY:
A thorough characterization of glucose metabolism and "inflammaging" in elderly subjects will help determine to what extent each of these factors affects muscle mass/function and contributes to age-related muscle wasting. The investigators will correlate patterns of insulin secretion/sensitivity with "muscle "quality/quantity" in diabetic and non-diabetic elderlies (≥70 years old). By comparing different groups (healthy, sarcopenic, diabetic, diabetic/sarcopenic), the investigators expect to identify an "oxidative/inflammatory signature" (e.g., circulating interleukins/myokines, plasma antioxidant capacity) specific for the sarcopenic phenotype and related to muscle insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus: patients taking drugs for diabetes will be diagnosed as having diabetes. In all other patients, a diagnosis will be established according to the criteria of the American Diabetes Association
* Sarcopenia (non-severe): individuals with low muscle mass and either low muscle strength or low physical performance will be diagnosed with sarcopenia, according to the criteria of the European Working Group on Sarcopenia in Older People (EWGSOP)
* Healthy volunteers: no diabetes, no sarcopenia and none of the exclusion criteria

Exclusion Criteria (overall population):

* acute diseases,
* chronic obstructive pulmonary disease (COPD)
* conditions associated with sarcopenia/altered body composition (e.g. disability, altered endocrine function, chronic diseases, nutritional deficiencies, cancer),
* obesity (body mass index ≥30 kg/m2)
* moderate-severe hepatic disease,
* chronic kidney disease (estimated glomerular filtration rate <30 ml/min per 1.73m2),
* metal prostheses,
* recent or ongoing infection,
* inability or unwillingness to provide informed consent

Exclusion Criteria (diabetic population):

* type 1 diabetes,
* hemoglobin A1c >8.5% (69 mmol/mol),
* basal-bolus insulin therapy,
* insulin pump therapy,
* proliferative diabetic retinopathy,
* diabetic foot.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly (≥ 70 years) subjects
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers (TNF-α, interleukin-1, interleukin-2, interleukin-6, RANKL, Myostatin and GDF11) | 2 years
  The primary objective of the study is to detect differences in inflammatory markers in the four groups

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Catholic University of Sacred Heart, Rome
  - Ospedale San Giovanni Calibita - Fatebenefratelli Isola Tiberina, Rome